CLINICAL TRIAL: NCT04766736
Title: Netrin-1 in Hepatocellular Carcinoma: Pathology, Preclinical Targeting, and Definition of Eligibility Criteria for Phase 1 Trials
Brief Title: Netrin-1 & Hepatocellular Carcinoma HCC
Acronym: HCC-Net
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0258
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: HCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tumors (T) samples of various etiologies (HBV, HCV, NASH, alcool): The combination of the Tumors status of the sample combined with its etiology ((HBV, HCV, NASH, alcool)
  Interventions: Procedure: Quantification of netrin-1 signals by antibody-based approaches
- Non Tumors (NT) samples of various etiologies (HBV, HCV, NASH, alcool): The combination of the Non Tumors status of the sample combined with its etiology ((HBV, HCV, NASH, alcool)
  Interventions: Procedure: Quantification of netrin-1 signals by antibody-based approaches

INTERVENTIONS:
Procedure: Quantification of netrin-1 signals by antibody-based approaches — Samples have been obtained upon curative surgery without any other therapy administered and subsequently characterized by pathologists after FFPE inclusion.

SUMMARY:
Netrin-1 is a dependence receptor ligand participating in the pathology of several cancer types. It is up-regulated in chronic liver diseases, cirrhosis and HCC. We hypothesize that netrin-1 may play a detrimental role in HCC. The goal of this project is to characterize netrin-1 signals in HCC samples with ad hoc controls, to investigate the benefit of capturing netrin-1 in preclinical models of HCC and to try to define patients groups the most likely to benefit from this targeting approach in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* any patient suffering from HCC
* age >18
* informed consent provided

Exclusion Criteria:

- absence of informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both men and women, between 18 and 85 years of age, suffering from Hepatocellular Carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Netrin-1 expression patterns in HCC samples | Outcome measure is to be performed after surgery of the tumors (at least 1 year later). It has no impact on the patient's care.
  Netrin-1 expression levels will be quantified by immunoblotting with ad hoc internal standards. Positivity threshold by IHC will be evaluated using ad hoc positive and negative control tissues. The densitometry approach will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Hepatogastroenterology service of the Croix-Rousse Hospital, Lyon, France